CLINICAL TRIAL: NCT04563312
Title: Lower Limb Performance, Balance and Coordination Differences Between the Muay Thai Athletes and Recreational Bodybuilders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Cyprus International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-243
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Martial Arts; Body Building; Functional Performance
Keywords: Muay Thai; Body Building; Balance; Coordination; Lower Extremity Functional Performance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A total of 35 participants, 17 athletes (14 men and 3 women) engaged in MT and 18 athletes (13 men and 5 women) engaged in BB were included in the study
Masking Description: All the volunteers participating in the study signed the informed consent form and filled personal data forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Balance Assessment (No Intervention): The Flamingo Balance Test and Y Balance Test were used to evaluate static and dynamic balance, respectively.
- Coordination Assessment (No Intervention): Coordination was assessed using the Hexagon Test.
- Lower Extremity Functional Performance Assessment (No Intervention): Lower extremity functional performance was evaluated using the Single Leg Hop Test.
- Exercise (Experimental): Nine different clubs and sport centers were screened and 18- to 35-year-old individuals regularly engaged in MT or BB for the last 6 months were invited to join the study.
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — Nine different clubs and sport centers were screened and 18- to 35-year-old individuals regularly engaged in MT or BB for the last 6 months were invited to join the study.
  Arms: Exercise

SUMMARY:
Purpose: The aim of this study was to compare balance, coordination and lower extremity functional performances of Muay Thai (MT) athletes and bodybuilders (BB).

Method: Seventeen athletes (14 men and 3 women; mean age: 20.65 + 2.34) engaged in MT and 18 (13 men and 5 women, mean age: 25.89 + 4.83) engaged in BB were included in the study. The Flamingo Balance Test and Y Balance Test were used to evaluate static and dynamic balance, respectively. Coordination was assessed using the Hexagon Test. Lower extremity functional performance was evaluated using the Single Leg Hop Test.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-35 years
* Making MT and BB at least for 5 year as a professional athletes
* currently free of any lower limb injuries within the last three months
* no previous history of injury or surgery that may affect their lower limbs

Exclusion Criteria:

* trained less than 3 sessions per week
* having lower limb injury for more than 1 month
* having a history of surgery, or chronic and progressive disease in their lower limb
* having scoliosis or any other orthopaedic or neurological problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
The Flamingo Balance Test | 2 weeks
  The Flamingo Balance Test was used to evaluate static balance
Balance Assessment | 2 weeks
  The Y Balance Test was used to evaluate dynamic balance
Coordination Assessment | 2 weeks
  Coordination was assessed using the Hexagon Test
Lower Extremity Functional Performance Assessment | 2 weeks
  Lower extremity functional performance was evaluated using the Single Leg Hop Test.

CONTACTS AND LOCATIONS:
Overall Officials: Bünyamin Haksever, PhD, Study Director — Cyprus International University
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)